CLINICAL TRIAL: NCT00995059
Title: A Phase I/II Study of a Novel Reduced Intensity Conditioning Regimen for Allogeneic Stem Cell Transplantation in Patients With Multiple Myeloma
Brief Title: Bortezomib Before Donor Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC078F; NCI-2009-01249 (Registry Identifier: NCI-CTRP); 08-003029 (Other: Mayo Clinic IRB); MC078F (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Last update posted 2023-01-05 (Actual); Status verified 2011-02

CONDITIONS: Multiple Myeloma; Refractory Multiple Myeloma
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Transplantation; Bortezomib; Melphalan; Antilymphocyte Serum; thymoglobulin; Sirolimus; Tacrolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): CONDITIONING: Patients receive bortezomib IV and then undergo fractionated total-body irradiation on days -5 and -2. Patients receive thymoglobulin IV over 6 hours on days -5 to -2 and melphalan IV over 30 minutes on days -4 to -3. ALLOGENEIC STEM CELL TRANSPLANTATION: Patients undergo bone marrow or peripheral blood stem cell transplant on day 0. GRAFT-VS-HOST DISEASE PROPHYLAXIS: Beginning on day -3, patients receive oral sirolimus and taper beginning on day 61. Beginning on day -2, patients receive oral or IV tacrolimus and taper beginning on day 101.
  Interventions: Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: allogeneic bone marrow transplantation; Drug: bortezomib; Drug: melphalan; Drug: anti-thymocyte globulin; Drug: sirolimus; Drug: tacrolimus; Radiation: total-body irradiation

INTERVENTIONS:
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Undergo transplantation
Procedure: allogeneic bone marrow transplantation — Undergo transplantation
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; PS-341; VELCADE
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin; Melfalan
Drug: anti-thymocyte globulin — Given IV
  Other Names: ATG; ATGAM; lymphocyte immune globulin; Thymoglobulin
Drug: sirolimus — Given orally
  Other Names: AY 22989; RAPA; Rapamune; rapamycin; SILA 9268A; SLM
Drug: tacrolimus — Given oral or IV
  Other Names: Advagraf; FK 506; Prograf; Protopic
Radiation: total-body irradiation — Undergo total-body irradiation
  Other Names: TBI

SUMMARY:
Rationale: Giving bortezomib and low doses of chemotherapy and total-body irradiation before a donor stem cell transplant or peripheral blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving sirolimus and tacrolimus before and after transplant may stop this from happening.

Purpose: This phase I/II trial is studying the side effects and best dose of bortezomib before donor stem cell transplant in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
Objectives:

I. To determine the maximum tolerated dose (MTD) of bortezomib when used in a novel conditioning regimen for patients undergoing allogeneic stem cell transplantation for multiple myeloma.

II. To evaluate the tolerability and feasibility of this novel conditioning regimen and GVHD prophylaxis strategy incorporating several anti-myeloma agents, including bortezomib, in patients undergoing allogeneic stem cell transplantation for multiple myeloma.

III. To obtain an initial assessment of the efficacy of this novel conditioning regimen.

Outline: This is a phase I dose-escalation study of bortezomib followed by a phase II study.

Reduced-Intensity Conditioning: Patients receive bortezomib IV and then undergo fractionated total-body irradiation on days -5 and -2. Patients receive thymoglobulin IV over 6 hours on days -5 to -2 and melphalan IV over 30 minutes on days -4 to -3.

Allogenic Stem Cell Transplantation: Patients undergo bone marrow or peripheral blood stem cell transplant on day 0.

Graft versus Host Disease Prophylaxis: Beginning on day -3, patients receive oral sirolimus and taper beginning on day 61. Beginning on day -2, patients receive oral or IV tacrolimus and taper beginning on day 101. After completion of the study treatment, patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status (PS) 0, 1, or 2
* Diagnosis of symptomatic multiple myeloma
* High risk myeloma as defined by progressive disease =< 12 months after high dose chemotherapy and autologous HSC transplant or presences of poor prognostic features such as deletion of chromosome 13 or hypodiploidy by standard cytogenetics, or t(4; 14) by fluorescence in situ hybridization (FISH), or t(14;16) by FISH, or 17p- by FISH, or plasma cell labeling index >= 3%
* Availability of a HLA fully-matched or 1 mismatch related donor by low-resolution HLA typing for the loci A, B, C, DRB1 and DQB1 or HLA fully-matched unrelated donor by high-resolution typing for loci A, B, C and DRB1 and at least low-resolution for loci DQB1
* Recovery from toxicity of previous chemotherapy (excludes grade 1 neurotoxicity and hematological toxicity)
* Physically and psychologically capable of undergoing bone marrow or PBSC transplant
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control for the during of the study
* Male subject agrees to use an acceptable method for contraception for the duration of the study

Exclusion Criteria:

* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV hear failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* NOTE: Prior to study entry, and ECG abnormality at screening has to be documented by the investigator as not medically relevant
* Significant cardiac dysfunction defined as left ventricle ejection fraction < 40% or presence of symptomatic coronary artery disease
* Significant pulmonary disease defined as FEV < 50% or CLCO < 50% of the predicted values
* Pre existing peripheral neuropathy grade > 1
* Significant renal dysfunction defined as estimated creatinine clearance < 50 ml/min
* Significant liver dysfunction defined as total bilirubin >= 2 x upper limit of normal (ULN) or AST, ALT >= 3 x ULN
* Seroreactive for HIV, HTLV I or II, HBV, HCV
* Presence of uncontrolled bacterial, viral, or fungal infection
* Known allergy to any of the component of the investigational treatment regimen or required ancillary treatments
* Considered unable to tolerate the included doses of total body irradiation due to previous treatment with radiation
* Female subject is pregnant or breast-feeding
* Other active concurrent malignancy
* Prior allogeneic bone marrow/peripheral blood stem cell transplant
* Received other investigational drugs =< 14 days prior to enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Tolerability as assessed by CTCAE v3.0 (Phase I)
Assessment of toxicity (Phase I)
Proportion of successes
Transplant-related mortality (TRM) (Phase II) | 100 days
Rate acute graft-vs-host disease (GVHD) (Phase I)

SECONDARY OUTCOMES:
Rate of grades II-IV and grades III-IV acute graft-vs-host disease (GVHD)
Cumulative rate of chronic GVHD
Overall response
Overall survival
Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Martha Q. Lacy, M.D., Study Chair — Mayo Clinic; James L. Slack, M.D., Principal Investigator — Mayo Clinic